CLINICAL TRIAL: NCT06112561
Title: Fluctuation and Realbility of Cardiac Index and SVR/SVRI During Weaning From ECC Regarding Values Obtained From Femoral and Radial Artery Acumen IQ Sensor
Brief Title: Cardiac Index, SVR/SVRI During Weaning From ECC- Data Obtained From Femoral and Radial Artery Transducer
Acronym: RaFe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: George Papanicolaou Hospital (Other)
Responsible Party: Principal Investigator, Asouhidou Irene, Professor, George Papanicolaou Hospital
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: Aqumen23
Record Dates: First submitted 2023-10-22; First posted 2023-11-01 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Coronary Artery Disease; Aortic Valve Disease; Mitral Valve Disease
Keywords: cardiac output; cardiac index; systemic vascular resistance
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac output/index/SVR (Active Comparator): Record of CO/CI/SVR before and after weaning form ECC from radial and femoral artery cannula.
  Interventions: Device: CO/CI/SVR
- Hypotension event (Active Comparator): Prevent of hypotension event calculated from radial/femoral artery cannula
  Interventions: Device: CO/CI/SVR

INTERVENTIONS:
Device: CO/CI/SVR — fluctuations of CO/CI/SVR regarding data from radial or femoral arterial cannula, and the therapeutic intervention that it demands these values.

SUMMARY:
Swan Ganz catheter-Edwards Lifesciences obtains values of cardiac output/index and systemic vascular resistance/index using the mean artery pressure of either radial or femoral artery.

During weaning from extracorporeal circulation, arterial waveform-derived cardiac output measurements from radial cannulation site is not reliable as compared with measurements obtained from femoral cannulation site.

DETAILED DESCRIPTION:
50 consecutive cardiac surgical patients undergoing on-pump primary coronary artery bypass, valve replacement or combined surgery are included in the study. Cardiac output is measured sequentially by the arterial pressure waveform analysis method from radial and femoral arterial sites

ELIGIBILITY:
Inclusion Criteria: Coronary artery disease , aortic valve stenosis, aortic valve regurgitation, mitral valve stenosis, mitral valve regurgitation,

Exclusion Criteria: none

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Cardiac output | 5 minutes after weaning from extracorporeal circulation (ECC)
  Measurement of cardiac output from radial and femoral arterial cannula
Prediction of hypotension episode (HPI) | 5 minutes after weaning from ECC
  Measurement of possibility of hypotension episode (HPI) from femoral and radial arterial cannula
Systemic Vascular resistance (SVR) | 5 minutes after weaning from ECC
  Measurement of SVR from femoral and radial arterial cannula

CONTACTS AND LOCATIONS:
Overall Officials: Olga Ananiadou, MD,PhD, Study Chair — George PAPANIKOLAOU G.H.